CLINICAL TRIAL: NCT05072080
Title: A Phase 3 Safety, Immunogenicity, and Lot-Consistency Trial of the VLP-Based Chikungunya Vaccine PXVX0317 in Healthy Adults and Adolescents
Brief Title: A Phase 3 Trial of the VLP-Based Chikungunya Vaccine PXVX0317 (CHIKV VLP Vaccine)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EBSI-CV-317-004
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Results first posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Chikungunya Virus
Keywords: Chikungunya; VLP; PXVX0317; vaccine; immunogenicity; CHIKV
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 2:2:2:1 ratio within each age stratum (12 to <18, 18 to <46, and 46 to <65). This study will be conducted in the US, using up to 50 sites.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Group 1 - PXVX0317 lot A (Lot 104)
  Interventions: Biological: CHIKV VLP/adjuvant
- Group 2 (Experimental): Group 2 - PXVX0317 lot B (Lot 105)
  Interventions: Biological: CHIKV VLP/adjuvant
- Group 3 (Experimental): Group 3 - PXVX0317 lot C (Lot 106)
  Interventions: Biological: CHIKV VLP/adjuvant
- Group 4 (Placebo Comparator): Group 4 - Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CHIKV VLP/adjuvant — CHIKV VLP vaccine is comprised of chikungunya virus virus-like particles (CHIKV VLP), adsorbed on aluminum hydroxide adjuvant 2%
  Arms: Group 1; Group 2; Group 3
Biological: Placebo — Placebo is comprised of formulation buffer
  Arms: Group 4

SUMMARY:
The goal of this multi-center, randomized, double blind, placebo controlled study is to evaluate the safety and immunogenicity of PXVX0317 (CHIKV VLP vaccine) in healthy adult and adolescent subjects.

DETAILED DESCRIPTION:
Coprimary Objectives:

1. To evaluate the safety of PXVX0317 (CHIKV VLP vaccine) in healthy adult and adolescent participants 12 to <65 years of age.
2. To compare the anti-CHIKV serum neutralizing antibody (SNA) response to PXVX0317 (CHIKV VLP vaccine) and placebo at Day 22, as measured by geometric mean titer (GMT) and clinically relevant difference in seroresponse rate (PXVX0317 minus placebo).
3. To demonstrate the consistency of the anti-CHIKV SNA response across three consecutively manufactured lots of PXVX0317 (CHIKV VLP vaccine) at Day 22 as measured by GMT.

Secondary Objectives:

1. To compare the anti-CHIKV SNA response to PXVX0317 (CHIKV VLP vaccine) and placebo at Day 15, Day 183, and Day 8 as measured by GMT and seroresponse rate.
2. To compare the GMT fold increase in anti-CHIKV SNA response and number and percentage of participants with an anti-CHIKV SNA titer ≥15 and 4-fold rise over baseline, both at Day 8, 15, 22, and 183.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent (and assent, as applicable) voluntarily signed by participant (and guardian, as applicable).
* Males or females, 12 to <65 years of age.
* Generally healthy, in the opinion of the investigator, based on medical history, physical examination, and screening laboratory assessments.
* Women who are either: (i) Not of childbearing potential (CBP): pre-menarche, surgically sterile (at least six weeks post bilateral tubal ligation, bilateral oophorectomy or hysterectomy), or postmenopausal (defined as a history of ≥12 consecutive months without menses prior to randomization in the absence of other pathologic or physiologic causes, following cessation of exogenous sex-hormonal treatment) or (ii) Meeting all the below criteria: Negative serum pregnancy test at screening visit, Negative urine pregnancy test immediately prior to dosing at Day 1, Using an acceptable method of contraception (if women of CBP) for the duration of participation, such as hormonal contraceptives (eg, implants, pills, patches) initiated ≥30 days prior to dosing, intrauterine device (IUD) inserted ≥30 days prior to dosing, double barrier type of birth control (male condom with female diaphragm, male condom with cervical cap), Abstinence is acceptable only for adolescents (12 to <18 years old) who are not sexually active.

Exclusion Criteria:

* Currently pregnant, breastfeeding, or planning to become pregnant during the study.
* Body Mass Index (BMI) ≥35 kg/m2.
* Positive laboratory evidence of current infection with human immunodeficiency virus (HIV-1, HIV-2), hepatitis C virus (HCV) or hepatitis B virus (HBV).
* History of severe allergic reaction or anaphylaxis to any component of the vaccine.
* History of any known congenital or acquired immunodeficiency that could impact response to vaccination (eg, leukemia, lymphoma, generalized malignancy, functional or anatomic asplenia, alcoholic cirrhosis).
* Prior receipt or anticipated use of systemic immunomodulatory or immunosuppressive medications from six months prior to screening through Day 22. Note: For systemic corticosteroids, use at a dose or equivalent dose of 20 mg of prednisone daily for 14 days or more within three months of screening through Day 22 is exclusionary. The use of inhaled, intranasal, topical, ocular, or intraocular steroids is allowed.
* Receipt or anticipated receipt of blood or blood-derived products from 90 days prior to screening through Day 22.
* Acute disease within the last 14 days (participants with an acute mild febrile illness can be considered for a deferral of vaccination two weeks after the illness has resolved and treatment has been completed).
* Clinically significant cardiac, pulmonary, rheumatologic, or other chronic disease, in the opinion of the investigator. This may include chronic illness requiring hospitalization in the last 30 days prior to screening.
* Enrollment in an interventional study and/or receipt of another investigational product from 30 days prior to screening through the duration of study participation.
* Receipt or anticipated receipt of any vaccine from 30 days prior to Day 1 through Day 22.
* Evidence of substance abuse that, in the opinion of the investigator, could adversely impact the participant's participation or the conduct of the study.
* Prior receipt of an investigational CHIKV vaccine/product.
* Any other medical condition that, in the opinion of the investigator, could adversely impact the participant's participation or the conduct of the study.

Ages: 12 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3258 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Ajiboye, MD, Study Director — Bavarian Nordic
Locations (47):
- United States (47):
  - Optimal Research, LLC, Huntsville, Alabama
  - Alliance for Multispecialty Research - Mobile, Mobile, Alabama
  - Alliance for Multispecialty Research, LLC, Tempe, Arizona
  - Velocity Clinical Research, Banning, Banning, California
  - Optimal Research, LLC, San Diego, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Accel Research Sites-DeLand Clinical Research Unit, Lake Mary, Florida
  - Optimal Research, LLC, Melbourne, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Synexus Clinical Research US, Inc., Pinellas Park, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Velocity Clinical Research, Boise, Meridian, Idaho
  - Synexus Clinical Research US, Inc., Chicago, Illinois
  - Optimal Research LLC, Peoria, Illinois
  - Johnson County ClinTrials, Lenexa, Kansas
  - Alliance for Multispecialty Research, LLC, Newton, Kansas
  - Alliance for Multispecialty Research - Wichita East, Wichita, Kansas
  - Alliance for Multispecialty Research, LLC, Lexington, Kentucky
  - Alliance for Multispecialty Research, LLC, New Orleans, Louisiana
  - Optimal Research, LLC, Rockville, Maryland
  - Alliance for Multispecialty Research - Kansas City, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Synexus Clinical Research US, Inc., St Louis, Missouri
  - Wr-Crcn, Llc, Las Vegas, Nevada
  - Alliance for Multispecialty Research, LLC., Las Vegas, Nevada
  - Rochester Clinical Research, Inc., Rochester, New York
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Cincinnati Children's Hospital Medical Center - The Gamble Vaccine Research Center, Cincinnati, Ohio
  - Velocity Clinical Rsearch, Inc., Cleveland, Ohio
  - Aventiv Research Inc., Columbus, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Velocity Clinical Research, Medford, Medford, Oregon
  - Velocity Clinical Research-Providence, East Greenwich, Rhode Island
  - Synexus Clinical Research US, Inc., Anderson, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Velocity Clinical Research, Austin, Cedar Park, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Research Your Health, Plano, Texas
  - BFHC Research, San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - Alliance for Multispecialty Research, LLC, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Richardson JS, Anderson DM, Mendy J, Tindale LC, Muhammad S, Loreth T, Tredo SR, Warfield KL, Ramanathan R, Caso JT, Jenkins VA, Ajiboye P, Bedell L; EBSI-CV-317-004 Study Group. Chikungunya virus virus-like particle vaccine safety and immunogenicity in adolescents and adults in the USA: a phase 3, randomised, double-blind, placebo-controlled trial. Lancet. 2025 Apr 19;405(10487):1343-1352. doi: 10.1016/S0140-6736(25)00345-9. Epub 2025 Mar 27. PMID 40158526
- [Derived] Miao Q, Nguyen W, Zhu J, Liu G, van Oers MM, Tang B, Yan K, Larcher T, Suhrbier A, Pijlman GP. A getah virus-like-particle vaccine provides complete protection from viremia and arthritis in wild-type mice. Vaccine. 2024 Nov 14;42(25):126136. doi: 10.1016/j.vaccine.2024.07.037. Epub 2024 Jul 14. PMID 39004524
- [Derived] Bennett SR, McCarty JM, Ramanathan R, Mendy J, Richardson JS, Smith J, Alexander J, Ledgerwood JE, de Lame PA, Royalty Tredo S, Warfield KL, Bedell L. Safety and immunogenicity of PXVX0317, an aluminium hydroxide-adjuvanted chikungunya virus-like particle vaccine: a randomised, double-blind, parallel-group, phase 2 trial. Lancet Infect Dis. 2022 Sep;22(9):1343-1355. doi: 10.1016/S1473-3099(22)00226-2. Epub 2022 Jun 13. PMID 35709798

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted in the United States, using 47 sites. Healthy participants were enrolled in this study. Recruitment Period was from September 29, 2021 to October 06, 2022.
Groups:
- Group 1: Group 1 - PXVX0317 lot A
  CHIKV VLP/adjuvant: CHIKV VLP vaccine is comprised of chikungunya virus virus-like particles (CHIKV VLP), adsorbed on aluminum hydroxide adjuvant 2%
- Group 2: Group 2 - PXVX0317 lot B
  CHIKV VLP/adjuvant: CHIKV VLP vaccine is comprised of chikungunya virus virus-like particles (CHIKV VLP), adsorbed on aluminum hydroxide adjuvant 2%
- Group 3: Group 3 - PXVX0317 lot C
  CHIKV VLP/adjuvant: CHIKV VLP vaccine is comprised of chikungunya virus virus-like particles (CHIKV VLP), adsorbed on aluminum hydroxide adjuvant 2%
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 919 | 948 | 927 | 464
Completed | 803 | 837 | 832 | 430
Not Completed | 116 | 111 | 95 | 34
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 65 | 70 | 58 | 23
Not completed — Physician Decision | 2 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 45 | 30 | 27 | 7
Not completed — Sponsor Decision | 0 | 1 | 0 | 0
Not completed — Subject moved | 1 | 3 | 5 | 2
Not completed — Withdrawal by parent | 0 | 0 | 1 | 0
Not completed — Subject was deployed | 0 | 1 | 0 | 0
Not completed — Subject left site without receiving dose | 0 | 1 | 0 | 0
Not completed — Subject incarcerated | 0 | 1 | 0 | 1
Not completed — Noncompliance (protocol, study, visits, e-diary, etc.) | 0 | 2 | 1 | 1
Not completed — Subject missed last visit (Day 183) | 3 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Group 1 - PXVX0317 lot 104
  CHIKV VLP/adjuvant: CHIKV VLP vaccine is comprised of chikungunya virus virus-like particles (CHIKV VLP), adsorbed on aluminum hydroxide adjuvant 2%
- Group 2: Group 2 - PXVX0317 lot 105
  CHIKV VLP/adjuvant: CHIKV VLP vaccine is comprised of chikungunya virus virus-like particles (CHIKV VLP), adsorbed on aluminum hydroxide adjuvant 2%
- Group 3: Group 3 - PXVX0317 lot 106
  CHIKV VLP/adjuvant: CHIKV VLP vaccine is comprised of chikungunya virus virus-like particles (CHIKV VLP), adsorbed on aluminum hydroxide adjuvant 2%
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 919 | 948 | 927 | 464 | 3258
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (14.4) | 38 (14.3) | 39 (14.0) | 39 (14.4) | 39 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 452 | 506 | 478 | 231 | 1667
  Male | 467 | 442 | 449 | 233 | 1591
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 165 | 166 | 175 | 71 | 577
  Not Hispanic or Latino | 735 | 760 | 731 | 379 | 2605
  Unknown or Not Reported | 19 | 22 | 21 | 14 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 6 | 13 | 2 | 32
  Asian | 26 | 30 | 23 | 16 | 95
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 0 | 4 | 10
  Black or African American | 190 | 175 | 169 | 89 | 623
  White | 663 | 693 | 687 | 341 | 2384
  More than one race | 23 | 32 | 23 | 8 | 86
  Unknown or Not Reported | 4 | 8 | 12 | 4 | 28
Height [Mean (Standard Deviation); unit: cm] | 171.4 (10.03) | 170.4 (9.55) | 170.7 (10.02) | 171.2 (9.97) | 170.9 (9.89)
Weight [Mean (Standard Deviation); unit: kg] | 78.5 (16.50) | 78.4 (16.08) | 78.3 (16.42) | 77.6 (16.42) | 78.3 (16.34)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.63 (4.579) | 26.89 (4.480) | 26.73 (4.499) | 26.38 (4.570) | 26.70 (4.527)
Baseline Anti-CHIKV SNA Serostatus [Count of Participants; unit: Participants]
  Negative (<LLOQ) | 894 | 925 | 906 | 458 | 3183
  Positive (>=LLOQ) | 24 | 18 | 21 | 6 | 69
  Missing | 1 | 5 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Solicited Adverse Events (AE)
Description: Incidence of solicited AEs through Day 8 for PXVX0317 (CHIKV VLP vaccine) and placebo for all age strata combined (safety population).
Time Frame: 7 days post-vaccination
Population: The number of participants assessed is the number of safety population participants who completed a memory aid following the vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 906 | 939 | 920 | 458
Participants | 319 | 373 | 366 | 124

2. Primary Outcome: Incidence of Unsolicited AEs
Description: Incidence of unsolicited AEs through Day 29 for PXVX0317 (CHIKV VLP vaccine) and placebo for all age strata combined (safety population).
Time Frame: 28 days post-vaccination
Population: Safety population (vaccinated participants who provided safety assessment data), All ages pooled
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 918 | 945 | 927 | 464
Participants | 139 | 146 | 155 | 62

3. Primary Outcome: Incidence of Adverse Events of Special Interest (AESI)
Description: Incidence of AESIs, through Day 183 for PXVX0317 (CHIKV VLP vaccine) and placebo for all age strata combined (safety population).
Time Frame: 182 days post-vaccination
Population: Safety population (vaccinated participants who provided safety assessment data), All ages pooled
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 918 | 945 | 927 | 464
Participants | 3 | 2 | 1 | 1

4. Primary Outcome: Incidence of Medically Attended Adverse Event (MAAE)
Description: Incidence of MAAEs through Day 183 for PXVX0317 (CHIKV VLP vaccine) and placebo for all age strata combined (safety population).
Time Frame: 182 days post-vaccination
Population: Safety population (vaccinated participants who provided safety assessment data), All ages pooled
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 918 | 945 | 927 | 464
Participants | 81 | 83 | 85 | 42

5. Primary Outcome: Incidence of Serious Adverse Event (SAE)
Description: Incidence of SAEs through Day 183 for PXVX0317 (CHIKV VLP vaccine) and placebo for all age strata combined (safety population).
Time Frame: 182 days post-vaccination
Population: Safety population (vaccinated participants who provided safety assessment data), All ages pooled
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 918 | 945 | 927 | 464
Participants | 10 | 7 | 6 | 1

6. Primary Outcome: Anti-CHIKV Serum Neutralizing Antibody (SNA) Seroresponse Rates at Day 22
Description: Anti-CHIKV SNA seroresponse rates for PXVX0317 (CHIKV VLP vaccine) and placebo, difference (PXVX0317 minus placebo), and associated 95% confidence interval (CI) at Day 22 for the immunogenicity evaluable population (IEP), all age strata combined.
Time Frame: 21 days post-vaccination
Population: Immunogenicity evaluable population (randomized and vaccinated participants who provided an evaluable Day 22 anti-CHIKV SNA sample within the analysis window, had no measurable anti-CHIKV SNA titer at Day 1, and had no reason to be excluded as defined prior to unblinding). Groups 1, 2, and 3 are combined, as participants received same treatment of PXVX0317 (dose, adjuvant, schedule), with only difference being the lot of manufactured vaccine. Data is reported for PXVX0317 vaccinated vs. placebo.
Measure: Number (95% Confidence Interval); unit: percentage of participants (rounded)
Groups:
- PXVX0317: All participants that received active PXVX0317 vaccine, regardless of the manufactured vaccine lot. This includes all participants contained in Group 1, Group 2, and Group 3.
  CHIKV VLP/adjuvant: CHIKV VLP vaccine is comprised of chikungunya virus virus-like particles (CHIKV VLP), adsorbed on aluminum hydroxide adjuvant 2%
- Placebo: Group 4 - Placebo
  Placebo: Placebo is comprised of formulation buffer
Arm/Group | PXVX0317 | Placebo
Number analyzed (Participants) | 2559 | 424
percentage of participants (rounded) | 97.81 [97.2 to 98.3] | 1.18 [0.5 to 2.7]
Statistical Analysis 1: Comparison: PXVX0317 vs Placebo; Day 22; Test type: Superiority; p < 0.0001, Chi-squared — p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups. All 3 coprimary endpoints were required to be met for success, so no multiple comparisons were performed; Mean Difference (Final Values) = 96.6, 95% CI 2-sided [95.0 to 97.5] — Seroresponse rate difference is (PXVX0317 minus placebo)

7. Primary Outcome: Anti-CHIKV Serum Neutralizing Antibody (SNA) Seroresponse Rates at Day 22 (Data Reported Per Arm)
Description: Anti-CHIKV SNA seroresponse rates and associated 95% confidence interval for PXVX0317 (CHIKV VLP vaccine) and placebo at Day 22 for the immunogenicity evaluable population (IEP), all age strata combined.
Time Frame: 21 days post-vaccination
Population: Immunogenicity evaluable population (randomized and vaccinated participants who provided an evaluable Day 22 anti-CHIKV SNA sample within the analysis window, had no measurable anti-CHIKV SNA titer at Day 1, and had no reason to be excluded as defined prior to unblinding).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 841 | 860 | 858
percentage of participants | 98.1 [96.9 to 98.8] | 98.0 [96.9 to 98.8] | 97.3 [96.0 to 98.2]

8. Primary Outcome: Anti-CHIKV SNA Geometric Mean Titers (GMT) at Day 22
Description: Anti-CHIKV SNA GMTs and associated 95% CIs at Day 22 for PXVX0317 (CHIKV VLP vaccine) and placebo for the IEP, all age strata combined.
Time Frame: 21 days post-vaccination
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | PXVX0317 | Placebo
Number analyzed (Participants) | 2559 | 424
Titer | 1618 [1522 to 1720] | 8 [7 to 9]
Statistical Analysis 1: Comparison: PXVX0317 vs Placebo; Day 22; Test type: Superiority; p < 0.0001, ANOVA — All 3 coprimary endpoints were required to be met for success, so no multiple comparisons were performed; ANOVA model includes site and treatment group as fixed effects, assuming normality of log titers. p-value tests equivalence of group GMTs on log scale; GMT Ratio = 206, 95% CI 2-sided [183 to 232] — Ratio of GMTs is (PXVX0317:placebo)

9. Primary Outcome: Anti-CHIKV SNA Geometric Mean Titers (GMT) at Day 22 (Data Reported Per Arm - All Age Strata)
Description: as for outcome 8
Time Frame: 21 days post-vaccination
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 841 | 860 | 858
Titer | 1592 [1458 to 1739] | 1640 [1503 to 1789] | 1622 [1486 to 1771]

10. Primary Outcome: Anti-CHIKV SNA Geometric Mean Titers (GMT) at Day 22 (for Lot Comparison)
Description: Anti-CHIKV SNA GMTs and associated 95% CIs between all three pairs of PXVX0317 (CHIKV VLP vaccine) lots (104:105, 104:106, 105:106) in adults 18 to <46 years of age in the IEP at Day 22. Placebo group 4 is not relevant for this lot-to-lot consistency analysis.
  Reported GMT estimates and 95% CIs are derived from an ANOVA model that includes site and product lot as fixed effects assuming normality of log titers.
Time Frame: 21 days post-vaccination
Population: Adults 18 to <46 years in Immunogenicity evaluable population (randomized and vaccinated participants who provided an evaluable Day 22 anti-CHIKV SNA sample within the analysis window, had no measurable anti-CHIKV SNA titer at Day 1, and had no reason to be excluded as defined prior to unblinding). Placebo group 4 does not apply for this PXVX0317 lot-to-lot consistency analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 488 | 498 | 494
titer | 1857 [1641 to 2101] | 1887 [1672 to 2130] | 1950 [1724 to 2207]
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Equivalence — Success criterion was pairwise GMT ratios (104:105, 105:106, 104:106) each with a two-sided 95% CI within [0.667; 1.5]; GMT Ratio = 0.98, 95% CI 2-sided [0.85 to 1.14] — All 3 coprimary endpoints were required to be met for success, so no multiple comparisons were performed. GMT estimates and 95% CIs are derived from an ANOVA model that includes site and product lot as fixed effects assuming normality of log titers
Statistical Analysis 2: Comparison: Group 2 vs Group 3; Test type: Equivalence — Success criterion was pairwise GMT ratios (104:105, 105:106, 104:106) each with a two-sided 95% CI within [0.667; 1.5]; GMT Ratio = 0.97, 95% CI 2-sided [0.84 to 1.12] — [estimate comment as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: Group 1 vs Group 3; Test type: Equivalence — Success criterion was pairwise GMT ratios (104:105, 105:106, 104:106) each with a two-sided 95% CI within [0.667; 1.5]; GMT Ratio = 0.95, 95% CI 2-sided [0.82 to 1.10] — [estimate comment as in outcome 10, analysis 1]

11. Primary Outcome: Anti-CHIKV SNA Geometric Mean Titers (GMT) at Day 22 (Data Reported Per Arm - Adults 18 to <46)
Description: Anti-CHIKV SNA GMTs and associated 95% CIs for PXVX0317 (CHIKV VLP vaccine) and placebo in adults 18 to <46 years of age in the IEP at Day 22.
Time Frame: 21 days post-vaccination
Population: Adults 18 to <46 years in Immunogenicity evaluable population (randomized and vaccinated participants who provided an evaluable Day 22 anti-CHIKV SNA sample within the analysis window, had no measurable anti-CHIKV SNA titer at Day 1, and had no reason to be excluded as defined prior to unblinding).
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 488 | 498 | 494 | 245
Titer | 1838 [1638 to 2063] | 1866 [1666 to 2089] | 1932 [1721 to 2169] | 8 [7 to 10]

12. Secondary Outcome: Anti-CHIKV SNA Seroresponse Rates at Days 15, 183, and 8
Description: Anti-CHIKV SNA seroresponse rates for PXVX0317 (CHIKV VLP vaccine) and placebo, difference (PXVX0317 minus placebo), and associated 95% CIs at Day 15, Day 183, and Day 8, in that order, for the IEP, all age strata combined.
  Number analyzed is number of participants with a sample result available at the indicated visit.
Time Frame: Day 15, 183, and 8 (14, 182, and 7 days post-vaccination, respectively)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PXVX0317 | Placebo
Number analyzed (Participants) | 2559 | 424
percentage of participants
  Day 15: number analyzed (Participants) | 2434 | 395
  Day 15 | 96.8 [96.0 to 97.4] | 0.8 [0.3 to 2.2]
  Day 183: number analyzed (Participants) | 2301 | 401
  Day 183 | 85.5 [84.0 to 86.9] | 1.5 [0.7 to 3.2]
  Day 8: number analyzed (Participants) | 2510 | 419
  Day 8 | 46.6 [44.6 to 48.5] | 0.5 [0.1 to 1.7]
Statistical Analysis 1: Comparison: PXVX0317 vs Placebo; Day 15; Test type: Superiority; p < 0.0001, Chi-squared — Key secondary endpoints were tested hierarchically, such that each was only tested if all 3 coprimary endpoints and prior key secondary endpoints were met, so no multiple comparisons were performed; p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Mean Difference (Final Values) = 96.0, 95% CI 2-sided [94.3 to 96.8] — Seroresponse rate difference is (PXVX0317 minus placebo)
Statistical Analysis 2: Comparison: PXVX0317 vs Placebo; Day 183; Test type: Superiority; p < 0.0001, Chi-squared — [p-value comment as in outcome 12, analysis 1]; p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Mean Difference (Final Values) = 84.0, 95% CI 2-sided [81.7 to 85.6] — Seroresponse rate difference is (PXVX0317 minus placebo)
Statistical Analysis 3: Comparison: PXVX0317 vs Placebo; Day 8; Test type: Superiority; p < 0.0001, Chi-squared — [p-value comment as in outcome 12, analysis 1]; p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Mean Difference (Final Values) = 46.1, 95% CI 2-sided [43.8 to 48.1] — Seroresponse rate difference is (PXVX0317 minus placebo)

13. Secondary Outcome: Anti-CHIKV SNA Seroresponse Rates at Days 15, 183, and 8 (Data Reported Per Arm)
Description: Anti-CHIKV SNA seroresponse rates and associated 95% CIs for PXVX0317 (CHIKV VLP vaccine) and placebo at Day 15, Day 183, and Day 8, in that order, for the IEP, all age strata combined.
  Number analyzed is number of participants with a sample result available at the indicated visit.
Time Frame: Day 15, 183, and 8 (14, 182, and 7 days post-vaccination, respectively)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 841 | 860 | 858 | 424
percentage of participants
  Day 15: number analyzed (Participants) | 800 | 828 | 806 | 395
  Day 15 | 96.6 [95.1 to 97.7] | 97.1 [95.7 to 98.0] | 96.5 [95.0 to 97.6] | 0.8 [0.3 to 2.2]
  Day 183: number analyzed (Participants) | 752 | 772 | 777 | 401
  Day 183 | 84.6 [81.8 to 87.0] | 85.9 [83.2 to 88.2] | 86.0 [83.4 to 88.2] | 1.5 [0.7 to 3.2]
  Day 8: number analyzed (Participants) | 827 | 848 | 835 | 419
  Day 8 | 45.8 [42.5 to 49.2] | 47.8 [44.4 to 51.1] | 46.1 [42.8 to 49.5] | 0.5 [0.1 to 1.7]

14. Secondary Outcome: Anti-CHIKV SNA Geometric Mean Titers (GMTs) at Days 8, 15, and 183
Description: Anti-CHIKV SNA GMTs with associated 95% CIs at Day 8, Day 15, and Day 183 for PXVX0317 (CHIKV VLP vaccine) and placebo for the IEP, all age strata combined.
  Number analyzed is number of participants with a sample result available at the indicated visit.
Time Frame: Day 8, 15, and 183 (7, 14, and 182 days post-vaccination, respectively)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | PXVX0317 | Placebo
Number analyzed (Participants) | 2559 | 424
Titer
  Day 8: number analyzed (Participants) | 2510 | 419
  Day 8 | 93 [87 to 100] | 7 [6 to 8]
  Day 15: number analyzed (Participants) | 2434 | 395
  Day 15 | 1096 [1029 to 1167] | 8 [7 to 9]
  Day 183: number analyzed (Participants) | 2301 | 401
  Day 183 | 338 [318 to 358] | 8 [7 to 9]
Statistical Analysis 1: Comparison: PXVX0317 vs Placebo; Day 8; Test type: Superiority; p < 0.0001, ANOVA; [statistical method as in outcome 8, analysis 1]; GMT Ratio = 13, 95% CI 2-sided [11 to 14] — Ratio of GMTs is (PXVX0317:placebo)
Statistical Analysis 2: Comparison: PXVX0317 vs Placebo; Day 15; Test type: Superiority; p < 0.0001, ANOVA; [statistical method as in outcome 8, analysis 1]; GMT Ratio = 144, 95% CI 2-sided [128 to 162] — Ratio of GMTs is (PXVX0317:placebo)
Statistical Analysis 3: Comparison: PXVX0317 vs Placebo; Day 183; Test type: Superiority; p < 0.0001, ANOVA; [statistical method as in outcome 8, analysis 1]; GMT Ratio = 41, 95% CI 2-sided [37 to 46] — Ratio of GMTs is (PXVX0317:placebo)

15. Secondary Outcome: Anti-CHIKV SNA Geometric Mean Titers (GMTs) at Days 8, 15, and 183 (Data Reported Per Arm)
Description: as for outcome 14
Time Frame: Day 8, 15, and 183 (7, 14, and 182 days post-vaccination, respectively)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 841 | 860 | 858
Titer
  Day 8: number analyzed (Participants) | 827 | 848 | 835
  Day 8 | 90 [82 to 99] | 97 [88 to 106] | 93 [85 to 103]
  Day 15: number analyzed (Participants) | 800 | 828 | 806
  Day 15 | 1073 [981 to 1173] | 1112 [1019 to 1215] | 1102 [1007 to 1206]
  Day 183: number analyzed (Participants) | 752 | 772 | 777
  Day 183 | 331 [304 to 360] | 342 [315 to 372] | 340 [313 to 370]

16. Secondary Outcome: Geometric Mean Fold Increase (GMFI) in Anti-CHIKV SNA Titers From Day 1 to Days 8, 15, 22, and 183
Description: Geometric mean fold increase (GMFI) in anti-CHIKV SNA titers from Day 1 to Day 8, Day 15, Day 22, and Day 183 for the IEP for all age strata combined.
  Fold rise in geometric mean titer is the ratio of the post-baseline value to the baseline value (e.g. number of 2 represents a post-baseline doubling of geometric mean titer).
  Number analyzed is number of participants with a sample result available at both Day 1 and the indicated visit.
Time Frame: Day 8, 15, 22, and 183 (7,14, 21, and 182 days post-vaccination, respectively)
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise from baseline
Arm/Group | PXVX0317 | Placebo
Number analyzed (Participants) | 2559 | 424
Fold rise from baseline
  Day 8: number analyzed (Participants) | 2510 | 419
  Day 8 | 12.5 [11.6 to 13.3] | 1.0 [0.9 to 1.1]
  Day 15: number analyzed (Participants) | 2434 | 395
  Day 15 | 146.1 [137.2 to 155.6] | 1.0 [0.9 to 1.1]
  Day 22 | 215.7 [203.0 to 229.3] | 1.1 [0.9 to 1.2]
  Day 183: number analyzed (Participants) | 2301 | 401
  Day 183 | 45.0 [42.4 to 47.8] | 1.1 [1.0 to 1.2]
Statistical Analysis 1: Comparison: PXVX0317 vs Placebo; Day 8; Test type: Superiority; p < 0.0001, t-test, 2 sided — GMFI estimates and 95% CIs are based on t-statistics assuming a normal distribution of the log fold increase in titer. p-value tests equality of log fold increase in titer between groups
Statistical Analysis 2: Comparison: PXVX0317 vs Placebo; Day 15; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 3: Comparison: PXVX0317 vs Placebo; Day 22; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 16, analysis 1]
Statistical Analysis 4: Comparison: PXVX0317 vs Placebo; Day 183; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 16, analysis 1]

17. Secondary Outcome: Geometric Mean Fold Increase (GMFI) in Anti-CHIKV SNA Titers From Day 1 to Days 8, 15, 22, and 183 (Data Reported Per Arm)
Description: as for outcome 16
Time Frame: Day 8, 15, 22, and 183 (7,14, 21, and 182 days post-vaccination, respectively)
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise from baseline
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 841 | 860 | 858
Fold rise from baseline
  Day 8: number analyzed (Participants) | 827 | 848 | 835
  Day 8 | 12.0 [10.9 to 13.3] | 12.9 [11.7 to 14.2] | 12.5 [11.3 to 13.8]
  Day 15: number analyzed (Participants) | 800 | 828 | 806
  Day 15 | 143.1 [130.8 to 156.5] | 148.3 [135.7 to 162.0] | 147.0 [134.3 to 160.8]
  Day 22 | 212.3 [194.4 to 231.8] | 218.6 [200.4 to 238.6] | 216.3 [198.1 to 236.2]
  Day 183: number analyzed (Participants) | 752 | 772 | 777
  Day 183 | 44.1 [40.5 to 48.0] | 45.6 [41.9 to 49.6] | 45.4 [41.7 to 49.4]

18. Secondary Outcome: Number and Percentage of Participants With Anti-CHIKV SNA Titer ≥15 and 4-fold Rise Over Baseline at Days 8, 15, 22, and 183
Description: Number and percentage of participants with anti-CHIKV SNA titers ≥15 and 4-fold rise over baseline at Day 8, Day 15, Day 22, and Day 183 for the IEP for all age strata combined.
  Number analyzed is number of participants with a sample result available at the indicated visit.
Time Frame: Day 8, 15, 22, and 183 (7,14, 21, and 182 days post-vaccination, respectively)
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PXVX0317 | Placebo
Number analyzed (Participants) | 2559 | 424
percentage of participants
  SNA titers ≥15 at Day 8: number analyzed (Participants) | 2510 | 419
  SNA titers ≥15 at Day 8 | 91.9 [90.7 to 92.9] | 1.2 [0.5 to 2.8]
  SNA titers ≥15 at Day 15: number analyzed (Participants) | 2434 | 395
  SNA titers ≥15 at Day 15 | 99.5 [99.1 to 99.7] | 0.8 [0.3 to 2.2]
  SNA titers ≥15 at Day 22 | 99.2 [98.8 to 99.5] | 1.7 [0.8 to 3.4]
  SNA titers ≥15 at Day 183: number analyzed (Participants) | 2301 | 401
  SNA titers ≥15 at Day 183 | 99.0 [98.6 to 99.4] | 2.2 [1.2 to 4.2]
  ≥4-fold rise over baseline at Day 8: number analyzed (Participants) | 2510 | 419
  ≥4-fold rise over baseline at Day 8 | 65.5 [63.6 to 67.3] | 0.7 [0.2 to 2.1]
  ≥4-fold rise over baseline at Day 15: number analyzed (Participants) | 2434 | 395
  ≥4-fold rise over baseline at Day 15 | 98.6 [98.0 to 99.0] | 0.8 [0.3 to 2.2]
  ≥4-fold rise over baseline at Day 22 | 98.6 [98.1 to 99.0] | 1.4 [0.7 to 3.1]
  ≥4-fold rise over baseline at Day 183: number analyzed (Participants) | 2301 | 401
  ≥4-fold rise over baseline at Day 183 | 92.9 [91.8 to 93.9] | 1.5 [0.7 to 3.2]
Statistical Analysis 1: Comparison: PXVX0317 vs Placebo; SNA titers ≥15 at Day 8; Test type: Superiority; p < 0.0001, Chi-squared; p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Mean Difference (Final Values) = 90.7, 95% CI 2-sided [88.7 to 91.9] — Seroresponse rate difference is (PXVX0317 minus placebo)
Statistical Analysis 2: Comparison: PXVX0317 vs Placebo; SNA titers ≥15 at Day 15; Test type: Superiority; p < 0.0001, Chi-squared — p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Mean Difference (Final Values) = 98.7, 95% CI 2-sided [97.2 to 99.3] — Seroresponse rate difference is (PXVX0317 minus placebo)
Statistical Analysis 3: Comparison: PXVX0317 vs Placebo; SNA titers ≥15 at Day 22; Test type: Superiority; p < 0.0001, Chi-squared; p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Mean Difference (Final Values) = 97.6, 95% CI 2-sided [95.8 to 98.5] — Seroresponse rate difference is (PXVX0317 minus placebo)
Statistical Analysis 4: Comparison: PXVX0317 vs Placebo; SNA titers ≥15 at Day 183; Test type: Superiority; p < 0.0001, Chi-squared; p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Mean Difference (Final Values) = 96.8, 95% CI 2-sided [94.8 to 97.9] — Seroresponse rate difference is (PXVX0317 minus placebo)
Statistical Analysis 5: Comparison: PXVX0317 vs Placebo; ≥4-fold rise over baseline at Day 8; Test type: Superiority; p < 0.0001, Chi-squared; p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Mean Difference (Final Values) = 64.8, 95% CI 2-sided [62.5 to 66.7] — Seroresponse rate difference is (PXVX0317 minus placebo)
Statistical Analysis 6: Comparison: PXVX0317 vs Placebo; ≥4-fold rise over baseline at Day 15; Test type: Superiority; p < 0.0001, Chi-squared; p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Mean Difference (Final Values) = 97.8, 95% CI 2-sided [96.3 to 98.4] — Seroresponse rate difference is (PXVX0317 minus placebo)
Statistical Analysis 7: Comparison: PXVX0317 vs Placebo; ≥4-fold rise over baseline at Day 22; Test type: Superiority; p < 0.0001, Chi-squared; p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Mean Difference (Final Values) = 97.2, 95% CI 2-sided [95.5 to 98.1] — Seroresponse rate difference is (PXVX0317 minus placebo)
Statistical Analysis 8: Comparison: PXVX0317 vs Placebo; ≥4-fold rise over baseline at Day 183; Test type: Superiority; p < 0.0001, Chi-squared; p-value is from a two-sided chi-square test of equality of seroresponse percentages between groups; Mean Difference (Final Values) = 91.4, 95% CI 2-sided [89.4 to 92.7] — Seroresponse rate difference is (PXVX0317 minus placebo)

19. Secondary Outcome: Number and Percentage of Participants With Anti-CHIKV SNA Titer ≥15 and 4-fold Rise Over Baseline at Days 8, 15, 22, and 183 (Data Reported Per Arm)
Description: as for outcome 18
Time Frame: Day 8, 15, 22, and 183 (7,14, 21, and 182 days post-vaccination, respectively)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 841 | 860 | 858
percentage of participants
  SNA titers ≥15 at Day 8: number analyzed (Participants) | 827 | 848 | 835
  SNA titers ≥15 at Day 8 | 90.9 [88.8 to 92.7] | 93.6 [91.8 to 95.1] | 91.0 [88.9 to 92.8]
  SNA titers ≥15 at Day 15: number analyzed (Participants) | 800 | 828 | 806
  SNA titers ≥15 at Day 15 | 99.4 [98.5 to 99.7] | 99.5 [98.8 to 99.8] | 99.5 [98.7 to 99.8]
  SNA titers ≥15 at Day 22 | 99.3 [98.5 to 99.7] | 99.2 [98.3 to 99.6] | 99.2 [98.3 to 99.6]
  SNA titers ≥15 at Day 183: number analyzed (Participants) | 752 | 772 | 777
  SNA titers ≥15 at Day 183 | 98.9 [97.9 to 99.5] | 99.0 [98.0 to 99.5] | 99.2 [98.3 to 99.6]
  ≥4-fold rise over baseline at Day 8: number analyzed (Participants) | 827 | 848 | 835
  ≥4-fold rise over baseline at Day 8 | 66.7 [63.5 to 69.9] | 66.0 [62.8 to 69.1] | 63.7 [60.4 to 66.9]
  ≥4-fold rise over baseline at Day 15: number analyzed (Participants) | 800 | 828 | 806
  ≥4-fold rise over baseline at Day 15 | 98.1 [96.9 to 98.9] | 98.8 [97.8 to 99.3] | 98.8 [97.7 to 99.3]
  ≥4-fold rise over baseline at Day 22 | 98.7 [97.7 to 99.3] | 98.7 [97.7 to 99.3] | 98.5 [97.4 to 99.1]
  ≥4-fold rise over baseline at Day 183: number analyzed (Participants) | 752 | 772 | 777
  ≥4-fold rise over baseline at Day 183 | 92.0 [89.9 to 93.8] | 93.5 [91.6 to 95.1] | 93.2 [91.2 to 94.7]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 through to the Day 183 end of study visit.
Description: Solicited AE is a protocol-specified AE which is proactively asked of the participant during a protocol-specified time period (Systematic assessment).
  Unsolicited AE is spontaneously reported by participant or discovered by investigator (Non-systematic assessment).
Groups:
- Group 1 - PXVX0317 Lot 104; Group 2 - PXVX0317 Lot 105; Group 3 - PXVX0317 Lot 106: CHIKV VLP/adjuvant: CHIKV VLP vaccine is comprised of chikungunya virus virus-like particles (CHIKV VLP), adsorbed on aluminum hydroxide adjuvant 2%
- Group 4 - Placebo: Placebo: Placebo is comprised of formulation buffer
Arm/Group | Group 1 - PXVX0317 Lot 104 | Group 2 - PXVX0317 Lot 105 | Group 3 - PXVX0317 Lot 106 | Group 4 - Placebo
All-Cause Mortality (participants affected / at risk) | 0/918 | 0/945 | 1/927 | 0/464
Serious Adverse Events (participants affected / at risk) | 10/918 | 7/945 | 6/927 | 1/464
Other Adverse Events (participants affected / at risk) | 323/918 | 375/945 | 367/927 | 127/464
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - PXVX0317 Lot 104 (N=918) | Group 2 - PXVX0317 Lot 105 (N=945) | Group 3 - PXVX0317 Lot 106 (N=927) | Group 4 - Placebo (N=464)
Arnold-Chiari malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — single reported event was a pre-existing condition diagnosed during the study
Encephalocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal ganglia infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - PXVX0317 Lot 104 (N=918) | Group 2 - PXVX0317 Lot 105 (N=945) | Group 3 - PXVX0317 Lot 106 (N=927) | Group 4 - Placebo (N=464)
Nausea (Gastrointestinal disorders) | 64 (64) | 75 (79) | 73 (78) | 31 (31)
Injection site pain (General disorders) | 200 (200) | 234 (235) | 223 (226) | 49 (49)
Fatigue (General disorders) | 169 (171) | 198 (201) | 190 (192) | 79 (79)
Chills (General disorders) | 69 (69) | 79 (79) | 91 (92) | 15 (15)
Myalgia (Musculoskeletal and connective tissue disorders) | 151 (152) | 166 (167) | 171 (173) | 45 (46)
Arthralgia (Musculoskeletal and connective tissue disorders) | 63 (66) | 87 (88) | 75 (76) | 34 (36)
Headache (Nervous system disorders) | 146 (150) | 176 (180) | 186 (193) | 78 (78)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This is a multi-center study and agreements with investigators depends on the individual site contract.

DOCUMENTS (2):
  • Study Protocol (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT05072080/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/80/NCT05072080/SAP_001.pdf